CLINICAL TRIAL: NCT05046236
Title: Developing Visual Feedback-aided Power Rehabilitation System and Exploring Its' Applications on Rehabilitation Training for Patients With Parkinson's Disease
Brief Title: Interactive POWER Rehabilitation System on Rehabilitation Training for Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-05-004A
Record Dates: First submitted 2021-07-29; First posted 2021-09-16 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
Keywords: Interactive POWER rehabilitation; Applications; Data analysis; Laser sensors; Parkinson's disease; Machine learning; Physical function; Exercise intervention; Activities of daily living; Functional training; Quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive POWER rehabilitation (Experimental): Participants in this group would be treated with POWER for twice a week, total 12 weeks.
  Interventions: Other: Interactive POWER rehabilitation
- Conventical physical training Group (Active Comparator): Participants in this group would be treated with traditional exercise rehabilitation for twice a week, total 12 weeks.
  Interventions: Other: Conventical physical training
- Control group (No Intervention): Usual care

INTERVENTIONS:
Other: Interactive POWER rehabilitation — Interactive POWER rehabilitation training for twice a week, total 12 weeks, that consisted of 6 types of equipment for strength training.
  Arms: Interactive POWER rehabilitation
Other: Conventical physical training — Conventional physical training models in current clinical use for twice a week, total 12 weeks, that consisted of strength training, balance training, stretching, gait training, and etc.
  Arms: Conventical physical training Group

SUMMARY:
In the previous studies, progressive resistance training (PRT) has significantly improved the muscle strength and disease severity of Parkinson's disease. However, there is currently no consensus on the impact of PRT on physical function such as balance and walking ability for Parkinson's patients. Therefore, this study focuses on developing a visual feedback system added to the original POWER rehabilitation system, and to investigate whether the training through this "interactive POWER rehabilitation system" can produce the clinical benefits, as well as improving the daily life of patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disease of the central nervous system with complex etiology. This disease is related to the consumption of dopamine in the substantia nigra of the brain, and it is currently believed that the main factors of consumption of dopamine are (1) heredity (2) aging (3) environment.

At present, there are many rehabilitation treatments available for patients with Parkinson's disease, such as: progressive resistance training, yoga, Tai Chi, dancing, cognitive training, balance training, gait training, bicycle, and treadmill training, etc. During the recent years, the POWER rehabilitation system from Japan (Procedure Outcome Worthwhile for Elderly Rehabilitation, referred to as POWER rehabilitation) including six types of equipment for strengthening different body parts has been applied to frail elderly or neurological patients gradually.

Parkinson's patients are often considered to have major difficulties in responding to motion disturbances (inability to respond appropriately), leading to learning, insufficient attention and motivation problems. Therefore, maintenance of motivation and feedback on performance are key factors that affect the participation of exercises in patients with Parkinson's disease.

The application of virtual reality in patients with PD is becoming more and more effective. An integrated rehabilitation system can not only enable the clinicians to check the rehabilitation status during the treatment, but also provide feedbacks to the patient through the interactive visual feedback screen. For Parkinson's patients, providing visual feedback through virtual reality intervention may be of particular clinical value.

In the first phase of this study, a virtual reality-like visual feedback system will be developed and combined with the original "POWER rehabilitation system" to form the so-called "Interactive POWER Rehabilitation System", and then system verification will be carried out. In the second phase of this study, this newly developed system will be applied to the rehabilitation training for patients with Parkinson's disease, and to explore whether the combination of POWER rehabilitation with visual feedback can produce the clinical benefits, as well as improving the daily life of patients with PD. Patients will be randomly assigned into three groups: interactive POWER, functional training, and control group. Single blind data collection will be used. Patients will be evaluated at baseline and post 12-week interventions. Outcome measures will include mini-BESTest, Unified Parkinson's disease rating scale, muscle strength of upper and lower extremities, timed up and go, 6-minute walking test, gait, and Parkinson's disease questionnaire PDQ-39.

It is expected that the "Interactive POWER Rehabilitation System" can promote the learning ability of patients with Parkinson's disease by adding visual feedbacks and enhance the treatment effects. It also offer rehabilitation clinicians more treatment options, lower the administrative costs of supporting staffs, reduce commuting costs for the patients, and elevate patients' desire to comply with the treatment program.

ELIGIBILITY:
Inclusion Criteria of phase I study

1. Healthy Volunteer (can walk 15 meters independently or with assistive devices).
2. Aged 20-70 years old.
3. Mini-mental state examination (MMSE) points above 24.
4. Not familiar with POWER rehabilitation machines before this study.
5. Able to understand POWER rehabilitation training and test items.
6. Able to use smart devices and be willing to cooperate with pre-acceptance instructions.
7. Able to communicate in Mandarin or Taiwanese, and be able to clearly express uncomfortable feelings.
8. Willing to participate in this study after explanations, and sign the subject's informed consent.

Inclusion Criteria of phase II study

1. Diagnosed as Idiopathic Parkinsonism by Neurologist
2. PD stages of I-III according to the modified Hoehn and Yahr Scale
3. Aged 45-85 years old
4. Mini-mental state testing (MMSE) 24 points or more
5. Stable medication regimen for at least 2 weeks before the trial
6. Can walk 15 meters independently or with devices
7. Able to understand treatment and assessment
8. Able to understand and be willing to agree to the informed consent form

Exclusion Criteria of phase I study

1. People who do not use smart devices and are unwilling to cooperate with the pre-acceptance instructions.
2. Have severe hearing or vision impairments.
3. Pregnant or breast-feeding.
4. Any chronic condition that may cause safety concerns.
5. Having any diseases which are contraindications for exercise participation.
6. Muscle strength is affected by taking drugs.
7. Have been to the gym 6 months before participating in the study (e.g. aerobic exercise, resistance training).
8. Severe orthopedic diseases (unhealed fractures, severe joint destructions, and joints with fixed deformities, etc.).
9. Severe or unstable neurological or cardiopulmonary diseases (severe cases of stroke and myocardial infarction in the acute phase, arrhythmia or uncontrolled blood pressure, etc.).
10. Diagnosed with any mental illness (e.g., depression, psychosis or other mental illnesses)
11. Unwilling to participate in this research.

Exclusion Criteria of phase II study

1. Rheumatism
2. Cardiovascular diseases or respiratory diseases (e.g., angina pectoris, pulmonary embolism, etc.)
3. Severe or unstable neurological or orthopedic diseases.
4. Severe hearing or vision impairments
5. Diagnosed with any mental illness(e.g., depression, psychosis or other mental illnesses)
6. A history of epilepsy.
7. Pregnancy or pregnancy
8. Any uncontrolled disease.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Unified Parkinson's Disease Rating Scale at 12 weeks | Baseline and post-intervention at 12 weeks
  A comprehensive assessment of both motor and non-motor symptoms associated with Parkinson's. The Unified Parkinson's Disease Rating Scale is made up of 42 items. These items are divided into six sections which are separately "evaluation of mentation, behavior, and mood", "self-evaluation of the activities of daily life", "clinician-scored monitored motor evaluation", "complications of therapy", "Hoehn and Yahr staging of severity of Parkinson's disease" and "Schwab and England ADL scale".The evaluation score for the first item to the 39th item is 0 to 4 points. The evaluation score for the 40th to the 42th item is 0 to 1 points. The higher score meand the worse condition. The sum of all the items'score is the score of the scale. Higher Rating Scales'scores indicate severe symptoms.
Change from Baseline he Parkinson's Disease Questionnaire (PDQ-39) at 12 weeks | Baseline and post-intervention at 12 weeks
  The 39-point PDQ provides scores for each of the 8 scales: mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communications and bodily discomfort. It is used to assess the overall health-related quality of life profile of the individual questioned.
Change from Baseline the Mini-Mental State Exam (MMSE) at 12 weeks | Baseline and post-intervention at 12 weeks
  A widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age.
Change from Baseline the Timed Up and Go test (TUG) at 12 weeks | Baseline and post-intervention at 12 weeks
  A simple test used to assess a person's mobility and requires both static and dynamic balance.
  It measures the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.
Change from Baseline Mini-BESTest at 12 weeks | Baseline and post-intervention at 12 weeks
  The scale includes four items: (1) anticipatory balance, (2) reactive posture control, (3) sensory orientation, and (4) dynamic gait, A total of 14 measurement items, 2 points for each question, a total of 28 points.
Change from Baseline six minute walk test (6MWT) at 12 weeks | Baseline and post-intervention at 12 weeks
  Walk for six minutes at the subject's preferred speed and assistive devices. You can stop at any time in the middle. After the end, the walking distance will be recorded, and changes in heartbeat, blood pressure, blood oxygen saturation, dyspnea and fatigue will be monitored. It will also end at the end then evaluate the walking distance.
Change from Baseline muscle strength of upper limbs at 12 weeks | Baseline and post-intervention at 12 weeks
  Use a hand-grip dynamometer to test the grip strength. Both hands need to be measured twice individually, with a rest time of at least 30 seconds between the two.
Change from Baseline muscle strength of lower limbs at 12 weeks | Baseline and post-intervention at 12 weeks
  Use Micro FET3 instrument to measure knee joint extension and flexion; hip joint abduction and flexion muscle strength. Each muscle group needs to be tested twice, with a 30-second rest between the two, and two recordings Take the maximum value afterwards.
Change from Baseline gait Speed at 12 weeks | Baseline and post-intervention at 12 weeks
  The subjects were asked to wear an inertial sensor "Physilog®" (Gait Up, Lausanne, Switzerland) on each foot during a 10-meter walking test to collect gait data. Spatiotemporal gait parameters were calculated with the Gait Analysis Software provided by Gait Up, including the following lists. Stopwatch will also be employed by the operator to measure the walking time simultaneously.
  - Speed (m/s): Mean walking stride velocity of forward walking
Change from Baseline cadence at 12 weeks | Baseline and post-intervention at 12 weeks
  The subjects were asked to wear an inertial sensor "Physilog®" (Gait Up, Lausanne, Switzerland) on each foot during a 10-meter walking test to collect gait data. Spatiotemporal gait parameters were calculated with the Gait Analysis Software provided by Gait Up.
  - Cadence (step/minute): Number of steps in a minute
Change from Baseline stride length at 12 weeks | Baseline and post-intervention at 12 weeks
  The subjects were asked to wear an inertial sensor "Physilog®" (Gait Up, Lausanne, Switzerland) on each foot during a 10-meter walking test to collect gait data. Spatiotemporal gait parameters were calculated with the Gait Analysis Software provided by Gait Up.
  - Stride length (m): Distance between two consecutive footprints on the ground

CONTACTS AND LOCATIONS:
Overall Officials: Si-Huei Lee, PhD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (2):
- Taiwan (2):
  - Far Eastern memorial hospital, New Taipei City
  - Taipei Veterans General Hospital, New Taipei City

IPD SHARING:
Plan to Share IPD: No